CLINICAL TRIAL: NCT03498027
Title: Febrile Whole Blood Specimen Collection and Testing Protocol to Demonstrate Product Specificity for the Applied Biosystems™ Bacillus Anthracis Detection Kit
Brief Title: Febrile Whole Blood Specimen Collection and Testing
Status: Completed | Type: Observational
Sponsor: MRI Global (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: MRI-2017-004/5
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Febrile Infection; Anthrax
MeSH Terms: conditions — Anthrax

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Febrile Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Data Collection
  Interventions: Device: TaqMan Bacillus anthracis Detection Kit

INTERVENTIONS:
Device: TaqMan Bacillus anthracis Detection Kit — The TaqMan® Bacillus anthracis Detection Kit is composed of the Applied Biosystems® 7500 Fast Dx Real-Time PCR Instrument with SDS Software, secondary interpretative software, and lyophilized reagents for the detection of gene targets for B. anthracis. The test assay is a multiplexed assay targeting gene targets for B. anthracis, in addition to an internal positive control. Reagents are lyophilized as a fully formulated Mastermix and are stable at room temperature for up to two years. The kit is specifically designed for performing real-time PCR using the Applied Biosystems® 7500 Fast Dx Real-Time PCR Instrument with SDS Software , with nucleic acids extracted from clinical specimens using Qiagen's QIAamp® Blood Midi Kit manual extraction or Roche MagNAPure automated extraction methods.

SUMMARY:
Whole blood samples will be collected from febrile patients presenting with fever of unknown origin and flu-like syndromes. Collection sites will consent patients and collect one (1) 4 mL whole blood sample from adults and either (1) 2 mL pediatric whole blood sample or 0.5 mL whole blood sample collected in a micro collection container from pediatric patients from each patient enrolled into the study. Study site will test whole blood samples received from collection sites daily using the Applied Biosystems™ Bacillus anthracis Detection Kit. Data generated will demonstrate product specificity when testing febrile whole blood samples.

DETAILED DESCRIPTION:
Whole blood samples will be collected from febrile patients presenting with fever of unknown origin and flu-like syndromes. Collection sites will be advised of collection requirements specific to patient population with the goal of collecting samples form patient between the ages of 2-89 years of age. Samples collected will be de-identified and assigned a specific study number. Study numbers and labels will be provided to collection site by the study monitor. Samples must be shipped to MRIGlobal or designated study site on the day of collection.

Collection sites will consent patients and collect one (1) 4 mL whole blood sample from adults and either (1) 2 mL pediatric whole blood sample or 0.5 mL whole blood sample collected in a micro collection container from pediatric patients (anticoagulant: K2EDTA or defined alternative) from each patient enrolled into the study. Patients may not be enrolled in the study more than once. Patients considered for enrollment will be logged on an enrollment log. Log must be reviewed by the site prior to considering a patient for study enrollment to confirm enrollment status. Samples collected will be de-identified and assigned a specific study number. Study numbers and labels will be provided to collection site by the study monitor.

Study site will accept or reject samples based on shipping verification procedures and then process samples acceptable for testing within 24 hours of receipt. Sample testing must be performed in accordance with the Applied Biosystems™ Bacillus anthracis Detection Kit instructions for use.

At study start, study site will test whole blood samples received from collection sites daily (e.g. Tuesday, Wednesday, Thursday, and Friday) using the Applied Biosystems™ Bacillus anthracis Detection Kit. No reference testing will be required since the study is designed only to demonstrate product specificity. Samples are assumed to be negative for Bacillus anthracis. A minimum of 50, but likely 100 febrile whole blood samples will be tested at MRIGlobal.

Data generated will demonstrate product specificity when testing febrile whole blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Fever

Exclusion Criteria:

* None

Ages: 2 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion criteria to be documented on data form provided.
  * Fever of unknown origin
  * Flu like syndrome
  Age ranges of study participants is as follows:
  2-15 Years of age 15-21 Years of age 22-40 Years of age >40 Years of age
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Product Specificity | 1 day
  Data generated will demonstrate product specificity when testing whole blood samples.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Boca Biolistics, Tarpon Springs, Florida
  - New England Center for Clinical Research, Fall River, Massachusetts
  - Medical Research Network, Franklin, Massachusetts

IPD SHARING:
Plan to Share IPD: No